CLINICAL TRIAL: NCT04893538
Title: Prognostic Value Of Lymphocyte Count and Lymphocyte/ Monocyte Ratio in Patients With Hodgkin's Lymphoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tishreen University (Other)
Responsible Party: Sponsor
Other Study IDs: Lymphopenia and Hodgkin
Record Dates: First submitted 2021-05-06; First posted 2021-05-19 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Hodgkin Lymphoma
Keywords: Lymphocyte count; International Prognostic Score; Lymphocyte/monocyte Ratio; Prognosis
MeSH Terms: conditions — Hodgkin Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- A: First analysis: Patients with high Lymphocyte count Second analysis: Patients with low International Prognosis Score Third analysis: Patients with high Lymphocyte/monocyte ratio
  Interventions: Diagnostic Test: First analysis: Lymphocyte count > or = 1500 cells per microlitre, second analysis: IPS < 3 and third analysis: Lymphocyte/Monocyte ratio > or = 2.9
- B: First analysis: Patients with low Lymphocyte count Second analysis: Patients with high International Prognostic Score Third analysis: Patients with low Lymphocyte/monocyte ratio
  Interventions: Diagnostic Test: First analysis: Lymphocyte count < 1500 cells per microlitre, second analysis: IPS > or = 3 and third analysis: Lymphocyte/Monocyte ratio < 2.9

INTERVENTIONS:
Diagnostic Test: First analysis: Lymphocyte count > or = 1500 cells per microlitre, second analysis: IPS < 3 and third analysis: Lymphocyte/Monocyte ratio > or = 2.9 — Intravenous blood sampling from participants for complete blood count to obtain Lymphocyte count, Monocyte count and Lymphocyte/Monocyte Ratio and for plasma Albumin to obtain IPS
  Groups: A
Diagnostic Test: First analysis: Lymphocyte count < 1500 cells per microlitre, second analysis: IPS > or = 3 and third analysis: Lymphocyte/Monocyte ratio < 2.9 — Intravenous blood sampling from participants for complete blood count to obtain Lymphocyte count, Monocyte count and Lymphocyte/Monocyte Ratio and for plasma Albumin to obtain IPS
  Groups: B

SUMMARY:
This study is to assess the utility of using Absolute Lymphocyte count, Lymphocyte/Monocyte Ratio and International Prognostic Scote at diagnosis in Hodgkin's Lymphoma as a prognostic predictor of therapeutic response, overall survival and progression free survival

DETAILED DESCRIPTION:
Hodgkin's Lymphoma has a high cure rate even if patients do not complete their treatment, this proposes that some patients may experience overtreatment and that would have negative effects (such as cardiac toxicity, sterility, secondary malignancies...) which makes it imperative to search for prognostic predictor suitable for all stages of disease, knowing that the International Prognostic Score "IPS" is restricted to advanced stages of the disease.

Absolute Lymphocyte count reflects the immune status of the individuals. It has been shown that an individual's immune status controls the extent of his response treatment, overall survival and his progression free survival because of the role that Lymphocytes play in suppressing and eliminating tumor cells.

Tumor-Associated Macrophages "TAMs" have been shown to play a role in tumor growth and development. Also, it has been shown that an increase in peripheral Monocyte count is associated with an increase in TAMs, so that the Monocyte count may constitute an important prognostic predictor.

Combining the Lymphocyte count and the Monocyte count into one index may be better for estimating the prognosis.

The aim of this study is to determine the prognostic significance of Absolute Lymphocyte count "ALC", Lymphocyte/Monocyte Ratio "LMR" and International Prognostic Score "IPS" at the cut-off points: 1500 cells per microliter for ALC, 2.9 for LMR and Score=3 for IPS.

Investigators get these cut-off points by conducting a retrospective case-control study on previous patients in Oncology Center, Tishreen Hospital, Syria in 2020.

This study will be prospective cohort :

1. participants will be divided into two subgroups (patients have ALC >= 1500 cells per microliter and who have ALC < 1500 cells per microliter). Those two subgroups will be homogenized in terms of other prognostic factors using Propensity Score.
2. the same participants will be also divided into another two subgroups (who have IPS < 3 and who have IPS >=3) and Those two subgroups will be homogenized using Propensity Score.
3. Finally the same participants will be divided into two subgroups (who have LMR >= 2.9 and who have LMR < 2.9) and Those two subgroups will be homogenized as mentioned before.

Then Investigators will monitor the therapeutic response, overall survival and progression free survival for 18 months for each subgroup and compare these indexes to determine the effectiveness of each of them in each stage of the disease

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed patients with Hodgkin's Lymphoma who have not yet received treatment
* Ages over 16 years old
* Signed informed consent before registration in study

Exclusion Criteria:

* Patients who have already received treatment
* Patients with a previous history of malignancy
* Patients with autoimmune diseases
* Patients with primary immunodeficiency
* AIDS patients
* Patients with acute or chronic infections
* Patients treated with drugs that affect the result of the analysis (Corticosteroids, Immunosuppressants, Li)

Min Age: 15 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients newly diagnosed with Hodgkin's lymphoma at the Oncology Center of Tishreen University Hospital who have not yet received treatment
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-01-04 (Actual); Primary Completion 2022-06-21 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Therapeutic response | 6 months
  Achieve complete remission after completing the prescribed treatment plan
overall survival | 18 months
  The occurrence of death after acceptance to study
progression free survival | 18 months
  The occurrence of relapse after acceptance to study

CONTACTS AND LOCATIONS:
Overall Officials: FIRAS Hussain, Dr., Study Chair — Tishreen University; Suzan Samra, Dr., Study Director — Tishreen University; Hasan Khalil, Principal Investigator — Tishreen University
Locations (1):
- Tishreen University, Latakia, Syria

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Background] Hancock BW, Dunsmore IR, Swan HT. Lymphopenia: a bad prognostic factor in Hodgkin's disease. Scand J Haematol. 1982 Sep;29(3):193-9. PMID 7146822
- [Background] Hasenclever D, Diehl V. A prognostic score for advanced Hodgkin's disease. International Prognostic Factors Project on Advanced Hodgkin's Disease. N Engl J Med. 1998 Nov 19;339(21):1506-14. doi: 10.1056/NEJM199811193392104. PMID 9819449
- [Background] Ayoub JP, Palmer JL, Huh Y, Cabanillas F, Younes A. Therapeutic and prognostic implications of peripheral blood lymphopenia in patients with Hodgkin's disease. Leuk Lymphoma. 1999 Aug;34(5-6):519-27. doi: 10.3109/10428199909058479. PMID 10492075
- [Background] Porrata LF, Ristow K, Colgan JP, Habermann TM, Witzig TE, Inwards DJ, Ansell SM, Micallef IN, Johnston PB, Nowakowski GS, Thompson C, Markovic SN. Peripheral blood lymphocyte/monocyte ratio at diagnosis and survival in classical Hodgkin's lymphoma. Haematologica. 2012 Feb;97(2):262-9. doi: 10.3324/haematol.2011.050138. Epub 2011 Oct 11. PMID 21993683
- [Background] Koh YW, Kang HJ, Park C, Yoon DH, Kim S, Suh C, Go H, Kim JE, Kim CW, Huh J. The ratio of the absolute lymphocyte count to the absolute monocyte count is associated with prognosis in Hodgkin's lymphoma: correlation with tumor-associated macrophages. Oncologist. 2012;17(6):871-80. doi: 10.1634/theoncologist.2012-0034. Epub 2012 May 15. PMID 22588324
- [Background] Tadmor T, Polliack A. Lymphopenia a simple prognostic factor in lymphoma and other cancers: why not use it more as a guide? Leuk Lymphoma. 2010 Oct;51(10):1773-4. doi: 10.3109/10428194.2010.508825. No abstract available. PMID 20849382